CLINICAL TRIAL: NCT03563287
Title: Altered Metabolism of Nutrients and Drugs in Obesity and After Obesity Surgery
Brief Title: Effects of LRYGB on Pharmacokinetics of Nine CYP Probe Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Diabetes Research Foundation, Finland (Other); Finnish Cultural Foundation (Other); Kuopio University Hospital (Other); Academy of Finland (Other)
Responsible Party: Principal Investigator, Jussi Pihlajamäki, Prof., University of Eastern Finland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NUDROBE
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenotyping cocktail of 9 CYP probe drugs before surgery (Experimental)
  Interventions: Drug: cocktail of nine CYP probe drugs
- Phenotyping cocktail of 9 CYP probe drugs 1 year after surgery (Experimental)
  Interventions: Drug: cocktail of nine CYP probe drugs

INTERVENTIONS:
Drug: cocktail of nine CYP probe drugs — Two equally loaded capsules containing:
  Melatonin (2.0 mg) Nicotine (1.0 mg) Bupropion (37.5 mg) Repaglinide (0.25 mg) Losartan (12.5 mg) Omeprazole (10 mg) Chlorzoxazone (62.5 mg) Midazolam (1.85 mg) Dextromethorphan (30 mg) as an oral solution was administered separately after the capsules.

SUMMARY:
Due to anatomical and physiological changes caused by the Roux-en-Y gastric bypass (RYGB) bariatric surgery, drug bioavailability after the surgery can be altered. Therefore, post-operative dose adjustment in these patients can be required.

The aim of the study was to investigate the effects of laparoscopic Roux-en-Y gastric bypass (LRYGB) surgery on drug pharmacokinetics and cytochrome P450 (CYP) mediated metabolism using a cocktail of nine CYP probe drugs.

The cocktail covers nine main CYP enzymes: melatonin (CYP1A2), nicotine (CYP2A6), bupropion (CYP2B6), repaglinide (CYP2C8), losartan (CYP2C9), omeprazole (CYP2C19/CYP3A4), dextromethorphan (CYP2D6), chlorzoxazone (CYP2E1), midazolam (CYP3A4).

The changes in pharmacokinetic parameters of the drugs as well as modulation of the activity of CYPs are evaluated before and one year after LRYGB. In the study, the patients administering drug cocktail before surgery and 1 year after LRYGB are served as their own controls.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 kg/m2 or BMI 35-40 kg/m2 and a comorbidity or its risk factor, such as type 2 diabetes, hypertension, sleep apnea, osteoarthritis of weight bearing joints or polycystic ovarian syndrome;
* previous conservative treatment for obesity had been proven to be ineffective;
* patients were assigned to undergo LRYGB surgery
* patients are able to give a written inform consent.

Exclusion Criteria:

* smokers
* consuming alcohol more than 20 g per day were included in the study
* taking drugs which alter CYPs activity
* history of hypersensitivity to the drugs used in the cocktail

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-01-27 (Actual); Primary Completion 2014-12-10 (Actual); Study Completion 2014-12-10 (Actual)

PRIMARY OUTCOMES:
Probe cocktail drugs concentration-time profile in plasma and urine before LRYGB | baseline, 1 hour, 2 hour, 4 hour and 6 hour
Probe cocktail drugs concentration-time profile in plasma and urine 1 year after LRYGB | baseline, 1 hour, 2 hour, 4 hour and 6 hour

SECONDARY OUTCOMES:
Metabolic ratios of parent compounds and corresponding metabolites before LRYGB | baseline, 1 hour, 2 hour, 4 hour and 6 hour
Metabolic ratios of parent compounds and corresponding metabolites 1 year after LRYGB | baseline, 1 hour, 2 hour, 4 hour and 6 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No